CLINICAL TRIAL: NCT06258798
Title: Comparison of the Dental X-ray Analysis Performed by an Artificial Intelligence Algorithm and the Analysis Performed by Dentists
Brief Title: The Use of Artificial Intelligence in the Dental X-rays Analysis
Status: Completed | Type: Observational
Sponsor: Hospital of the Ministry of Interior, Kielce, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: CT/2023/1
Record Dates: First submitted 2024-01-25; First posted 2024-02-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Oral Health; Dental Caries; Periapical Diseases; Tooth Loss
MeSH Terms: conditions — Dental Caries; Periapical Diseases; Tooth Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- One group of patients (double gate): Study design:
  * Direction of data collection: retrospective
  * Number of gates (sets of eligibility criteria): double gate (AI, human)
  * Participant sampling method: Consecutive
  * Method of allocating participants to index tests: Each participant received all index tests
  * Number of reference standards: Single test standard
  * Limited verification: Full verification (not limited)
  Interventions: Radiation: Taking a dental X-ray

INTERVENTIONS:
Radiation: Taking a dental X-ray — Dental X-rays taken in patients with indications confirmed by a written referral.

SUMMARY:
This cross-sectional study aims to perform a population-based assessment of the incidence of decay, dental fillings, root canal fillings, endodontic lesions, implants, implant and dental abutment crowns, pontic crowns, and missing teeth, taking into account the location.

DETAILED DESCRIPTION:
This cross-sectional study aims to perform a population-based assessment of the incidence of decay, dental fillings, root canal fillings, endodontic lesions, implants, implant and dental abutment crowns, pontic crowns, and missing teeth, considering the location. Patients with indications for dental X-ray confirmed by a written referral and with permanent dentition will participate in the study. Then, the X-rays will be analyzed by the dentists and the AI-based software after the data has been anonymized. The results will be compared to determine the AI algorithm's sensitivity, specificity, and precision.

ELIGIBILITY:
Inclusion Criteria:

* Indications for dental X-ray confirmed by a written referral from the dentist or physician (both screening tests and tests performed for treatment purposes were allowed)
* Permanent dentition (after exfoliation is completed)

Exclusion Criteria:

* Patients with mixed dentition (exfoliation has not finished)

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in the study were admitted to the radiology department in Kielce, a city in southern Poland with around 200.000 inhabitants.
Sampling Method: Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Up to 6 weeks
  Sensitivity (also known as recall or true positive rate) is the proportion of actual positive cases that are correctly predicted as positive. It evaluates the performance of an AI algorithm. Formally it can be calculated with the following equation:
  Sensitivity = TP / (TP+FN)
  True positive (TP) - a test result that correctly indicates the presence of a condition or characteristic
  False Negative (FN) - a test result which wrongly indicates that a particular condition or characteristic is absent
Specificity | Up to 6 weeks
  Specificity (also known as true negative rate) - is the proportion of actual negative cases that are correctly predicted as negative. It evaluates the performance of an AI algorithm. Formally it can be calculated by the equation below:
  Specificity = TN / (TN + FP)
  True negative (TN) - a test result that correctly indicates the absence of a condition or characteristic
  False positive (FP) - a test result which wrongly indicates that a particular condition or characteristic is present
Precision of the AI algorithm | Up to 6 weeks
  Precision is an evaluation metric used to assess the performance of machine learning algorithm for AI. It measures how accurate the algorithm is. We will use the number of true positives (TP) and false positives (FP) to calculate precision using the following formula:
  Precision = TP / (TP + FP)
  True positive (TP) - a test result that correctly indicates the presence of a condition or characteristic
  False positive (FP) - a test result that wrongly indicates that a particular condition or characteristic is present

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Sikora, Study Chair — Hospital of the Ministry of Interior, Wojska Polskiego 51, 25-375 Kielce, Poland
Locations (1):
- Department of Maxillofacial Surgery, Kielce, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turosz N, Checinska K, Checinski M, Lubecka K, Blizniak F, Sikora M. Artificial Intelligence (AI) Assessment of Pediatric Dental Panoramic Radiographs (DPRs): A Clinical Study. Pediatr Rep. 2024 Sep 11;16(3):794-805. doi: 10.3390/pediatric16030067. PMID 39311330